CLINICAL TRIAL: NCT02048176
Title: Long-Term Impact of Posterior Fossa Mutism on Quality of Life
Brief Title: Posterior Fossa Mutism on Quality of Life
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-14721
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2017-07

CONDITIONS: Posterior Fossa Mutism
Keywords: Mutism
MeSH Terms: conditions — Mutism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Posterior Fossa Mutism: Patients with Posterior Fossa Mutism
- Non Posterior Fossa Mutism: Patients that did not develop Mutism

SUMMARY:
Posterior fossa mutism (PFM) occurs in up to 30% of patients after resection of a posterior fossa tumor, most commonly a medulloblastoma. PFM is characterized by delayed onset of mutism 1-6 days after surgery that can spontaneously improve on average from 7-8 weeks later. Few patients recover normal speech. Most of their speech continues to be marked by dysarthria, dysfluency and slowed rate. Researchers have not identified the pathophysiologic mechanism for PFM nor have they found a cure. Despite the improvements in speech, patients with PFM have shown multiple areas of neurocognitive deficits 12 months after diagnosis. Few studies have looked at long term outcomes of patients affected by PFM. We propose to survey patients who developed PFM after resection of a medulloblastoma to determine long term effects of PFM on patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients must be between 8 years and 25 years of age at the time of enrollment and have completed treatment for their initial diagnosis of medulloblastoma.

Exclusion Criteria:

1. Patient is less than 8 years old or greater than 25 years old at the time of the administration of the survey.
2. Patients are too ill to complete the survey as identified by their treating physician.
3. Patients who are unable to speak or understand English.
4. Patients who are currently being treated for their original diagnosis of medulloblastoma.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients must be between 8 years and 25 years of age at the time of enrollment and have completed treatment for their initial diagnosis of medulloblastoma.
  We will identify a group of patients who developed PFM as well as a group of appropriately matched controls with regard to age, sex and treatment protocol who did not develop PFM.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Thirty minutes, no follow-up.

SECONDARY OUTCOMES:
quality of life in terms of anger, anxiety, depression, fatigue, social functioning, pain and stigma | 30 minutes, no follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gudrunardottir T, Sehested A, Juhler M, Schmiegelow K. Cerebellar mutism: review of the literature. Childs Nerv Syst. 2011 Mar;27(3):355-63. doi: 10.1007/s00381-010-1328-2. PMID 21061011
- [Background] Kupeli S, Yalcin B, Bilginer B, Akalan N, Haksal P, Buyukpamukcu M. Posterior fossa syndrome after posterior fossa surgery in children with brain tumors. Pediatr Blood Cancer. 2011 Feb;56(2):206-10. doi: 10.1002/pbc.22730. Epub 2010 Oct 25. PMID 21157890
- [Background] Palmer SL, Hassall T, Evankovich K, Mabbott DJ, Bonner M, Deluca C, Cohn R, Fisher MJ, Morris EB, Broniscer A, Gajjar A. Neurocognitive outcome 12 months following cerebellar mutism syndrome in pediatric patients with medulloblastoma. Neuro Oncol. 2010 Dec;12(12):1311-7. doi: 10.1093/neuonc/noq094. Epub 2010 Aug 16. PMID 20713408
- [Background] Szathmari A, Thiesse P, Galand-desme S, Mottolese C, Bret P, Jouanneau E, Guyotat J, Lion-Francois L, Frappaz D. Correlation between pre- or postoperative MRI findings and cerebellar sequelae in patients with medulloblastomas. Pediatr Blood Cancer. 2010 Dec 15;55(7):1310-6. doi: 10.1002/pbc.22802. PMID 20981689
- [Background] Wells EM, Walsh KS, Khademian ZP, Keating RF, Packer RJ. The cerebellar mutism syndrome and its relation to cerebellar cognitive function and the cerebellar cognitive affective disorder. Dev Disabil Res Rev. 2008;14(3):221-8. doi: 10.1002/ddrr.25. PMID 18924161
- [Background] Ozgur BM, Berberian J, Aryan HE, Meltzer HS, Levy ML. The pathophysiologic mechanism of cerebellar mutism. Surg Neurol. 2006 Jul;66(1):18-25. doi: 10.1016/j.surneu.2005.12.003. PMID 16793430
- [Background] Robertson PL, Muraszko KM, Holmes EJ, Sposto R, Packer RJ, Gajjar A, Dias MS, Allen JC; Children's Oncology Group. Incidence and severity of postoperative cerebellar mutism syndrome in children with medulloblastoma: a prospective study by the Children's Oncology Group. J Neurosurg. 2006 Dec;105(6 Suppl):444-51. doi: 10.3171/ped.2006.105.6.444. PMID 17184075